CLINICAL TRIAL: NCT00879203
Title: Glycemic Control, Brain Structure and Cognition in Youth With T1DM
Brief Title: Glycemic Control, Brain Structure and Cognition in Youth With Type 1 Diabetes (T1DM)
Acronym: LO5/HY5
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07-1258; R01DK064832-06 (NIH)
Record Dates: First submitted 2009-04-07; First posted 2009-04-09 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-10

CONDITIONS: Type 1 Diabetes Mellitis; Cognition
Keywords: Type 1 Diabetes Mellitis; Youth; Hypoglycemia; Hyperglycemia; Cognition; Memory; Brain Growth & Development; Magnetic Resonance Imaging
MeSH Terms: conditions — Hypoglycemia; Hyperglycemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Type 1 Diabetes (T1DM): Youth and young adults with T1DM
- Non diabetic siblings: Non diabetic, young siblings of T1DM participants

SUMMARY:
LO5 study: The investigators are inviting a new group of youth (ages 7-16) who have been recently diagnosed with type 1 diabetes and their non-diabetic siblings. These youth will complete cognitive tests and a MRI scan of the brain. This scan uses strong magnets to obtain pictures and does not involve any radiation or injections. The investigators will recruit patients within three months of their diagnosis date. The study entails 1 study visit that lasts 3.5 hours. Evening and weekend times are available. The investigators plan to enroll 135 participants.

HY5 study: The investigators are inviting a cohort of youth and young adults (ages 9-21) with type 1 diabetes and their non-diabetic siblings for a follow-up to a study they have already completed. This group of people will complete several memory and thinking tests along with several MRI scans of their brain, just as they did at their previous visits. The investigators plan to enroll 150 participants.

ELIGIBILITY:
LO5:

Inclusion Criteria for Participants with Type 1 Diabetes:

* Between the ages of 7 and 16
* Diagnosed with type 1 diabetes within 3 months

Inclusion Criteria for Participants without Type 1 Diabetes:

* Between the ages of 7 and 16

Exclusion Criteria for Participants with Type 1 Diabetes:

* Pregnant or lactating
* Chronic disease other than T1DM, well-controlled asthma, or Hashimoto's thyroiditis
* Other current serious medical illness
* Psychiatric illness
* Psychoactive drug dependence
* Neurological illness (except T1DM-related): stroke, seizure, major loss of consciousness, head injuries, encephalitis, or hydrocephalus, blindness, deafness
* Use of psychoactive medications or exposure to neuroleptics (except that exposures of less than 1 month, occurring more than 5 years ago, will be allowed)
* Use of dopamine depleting agents or stimulants such as Ritalin, Cylert, Adderall
* Pre-maturity at birth of more than 4 wks early with complications (e.g. on respirator at NICU)
* Inability to complete MRI scan (e.g. claustrophobia, metal implants)
* Full set (top and bottom) of orthodontic braces (Half set braces, fillings, and retainers are OK)

Exclusion Criteria for Participants without Type 1 Diabetes:

* Same as above (except cannot have type 1 diabetes)

HY5: Must have been a participant in our earlier study.

Ages: 7 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: LO5: Youth with type 1 diabetes (T1DM) between the ages of 7-16 who have been diagnosed within the previous 3 months. Non-diabetic siblings of the participants with T1DM aged 7-16 years old.
  HY5: Youth and young adults (ages 9-21) who have already completed an earlier study with the lab.
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2008-11; Primary Completion 2013-11 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara G. Hershey, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Perantie DC, Koller JM, Weaver PM, Lugar HM, Black KJ, White NH, Hershey T. Prospectively determined impact of type 1 diabetes on brain volume during development. Diabetes. 2011 Nov;60(11):3006-14. doi: 10.2337/db11-0589. Epub 2011 Sep 27. PMID 21953611